CLINICAL TRIAL: NCT00807105
Title: Evaluation of the H-coil Transcranial Magnetic Stimulation TMS Device - Safety and Feasibility Study for Acute and Maintenance Treatment in Major Depressive Episode
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shalvata Mental Health Center (Other)
Collaborators: Brainsway (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0013-07 SHA
Record Dates: First submitted 2008-11-20; First posted 2008-12-11 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Major Depressive Disorder
Keywords: MOOD EVALUATION
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- depressive patients (Experimental): patients suffering from deppresion
  Interventions: Device: H-coil dTMS

INTERVENTIONS:
Device: H-coil dTMS — treatment with deep TMS stimulation.

SUMMARY:
This is a prospective open label study of acute and maintenance treatment of MDD. The acute phase consists of daily treatments for 4 weeks. maintenance will be twice a week for eight weeks followed by 10 weeks of once a week treatments.

ELIGIBILITY:
Inclusion Criteria:

* MDD patients

Exclusion Criteria:

* risk factors for convulsions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
response in HAMDS | 1 YEAR

CONTACTS AND LOCATIONS:
Locations (1):
- ShalvataMHC, Hod HaSharon, Israel, Israel